CLINICAL TRIAL: NCT07218783
Title: A Prospective, Multicenter, Randomized, Masked, Controlled Study to Evaluate the Safety and Efficacy of the Bimatoprost Implant System (78 mcg) Used in Combination With the SpyGlass IOL Compared to Timolol Maleate Ophthalmic Solution, USP, 0.5%,
Brief Title: Evaluation of the Safety and Efficacy of the Bimatoprost Implant System Used in Combination With the SpyGlass IOL Compared to Timolol Ophthalmic Solution (Rhine)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: SpyGlass Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SGP-005
Record Dates: First submitted 2025-10-16; First posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Cataract; Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Cataract; Glaucoma; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bimatoprost Implant System / IOL Combination (Experimental)
  Interventions: Drug: Bimatoprost Implant System; Device: SpyGlass IOL
- Timolol Maleate Ophthalmic Solution 0.5% (Active Comparator)
  Interventions: Drug: Timolol Maleate Ophthalmic Solution, 0.5%; Device: Commercial IOL

INTERVENTIONS:
Drug: Bimatoprost Implant System — Bimatoprost Implant System used in combination with the SpyGlass IOL
  Arms: Bimatoprost Implant System / IOL Combination
Device: SpyGlass IOL — SpyGlass Intraocular Lens
  Arms: Bimatoprost Implant System / IOL Combination
Drug: Timolol Maleate Ophthalmic Solution, 0.5% — Timolol Maleate Ophthalmic Solution, 0.5% BID
  Arms: Timolol Maleate Ophthalmic Solution 0.5%
Device: Commercial IOL — Commercially Available Aspheric Monofocal Non-Yellow Chromophore Intraocular Lens
  Arms: Timolol Maleate Ophthalmic Solution 0.5%

SUMMARY:
This trial is a randomized study to evaluate the Bimatoprost Implant System used in combination with the SpyGlass IOL to Timolol Ophthalmic Solution in participants with mild to moderate open-angle glaucoma or ocular hypertension undergoing cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild to moderate open-angle glaucoma or ocular hypertension
* Planned removal of cataract
* Female participants of childbearing potential must have a negative urine pregnancy test at the baseline visit and agree to the use of contraception

Exclusion Criteria:

* Uncontrolled systemic disease
* History of incisional/refractive corneal surgery
* Any glaucoma diagnosis other than OHT, open-angle, pseudoexfoliative, or pigmentary glaucoma
* History of incisional glaucoma surgery or intraocular injections
* Other ocular diseases, pathology, or conditions

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
Mean IOP Reduction from Baseline (mmHg) | Weeks 2 and 6, and Month 3
  Time-matched mean IOP change from Baseline in the study eyes at all the individual IOP timepoints
BCDVA 20/40 or better | Month 6
  Study eyes achieving best corrected distance visual acuity (BCDVA) of 20/40 or better

SECONDARY OUTCOMES:
Mean IOP Reduction from Baseline (mmHg) | Month 6, 9 and 12
  Time matched mean IOP reduction from Baseline (mmHg) in the study eyes at all the individual IOP timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Paul Yoo, OD, Study Chair — SpyGlass Pharma
Locations (1):
- Houston Eye Associates, Houston, Texas, United States

REFERENCES:
- See also: SpyGlass Pharma Website — https://www.spyglasspharma.com/